CLINICAL TRIAL: NCT01137461
Title: Evaluation of Efficacy of Embryo Transfer Procedure Guided by Transvaginal Ultrasound Versus Abdominal Ultrasound in Recipients of Oocytes. A Single-centre, Randomized Clinical Trial.
Brief Title: Efficacy of Embryo Transfer Procedure Guided by Transvaginal Ultrasound Versus Abdominal Ultrasound in Oocytes Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Privada Eugin (Other)
Responsible Party: Dr. Daniel Bodri / Principal investigator, Clinica EUGIN
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TATV
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Infertility
Keywords: Female infertility with indication of oocyte reception
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- abdominal ultrasound (Other): traditional technique
  Interventions: Procedure: ultrasound-guided embryo transfer
- transvaginal ultrasound (Other): new technique
  Interventions: Procedure: ultrasound-guided embryo transfer

INTERVENTIONS:
Procedure: ultrasound-guided embryo transfer — Embryo transfer in oocyte recipients

SUMMARY:
The objective of this study is to evaluate the efficacy of embryo transfer procedure guided by transvaginal ultrasound versus abdominal ultrasound in recipients of oocytes as well as the advantages and disadvantages of the new technique.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte recipients.
* Uterus without previously detected anomalies.
* Patients able to understand the study requirements who want to participate during all its duration and that have signed the informed consent.

Exclusion Criteria:

* Turner syndrome, Black race (significantly lower implantational rates)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 40 days after embryo transfer
  Evidence of gestational sac by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bodri, Principal Investigator — Clinica EUGIN
Locations (1):
- Clinica EUGIN, Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Bodri D, Colodron M, Garcia D, Obradors A, Vernaeve V, Coll O. Transvaginal versus transabdominal ultrasound guidance for embryo transfer in donor oocyte recipients: a randomized clinical trial. Fertil Steril. 2011 Jun;95(7):2263-8, 2268.e1. doi: 10.1016/j.fertnstert.2011.03.028. Epub 2011 Apr 2. PMID 21459374
- See also: Clínica EUGIN — http://www.eugin.es/